CLINICAL TRIAL: NCT02523651
Title: Study of Local Periodontal Regeneration of Chronic Periodontal Disease Patients Receiving Allogeneic Human Dental Pulp Stem Cells Injection Therapy
Brief Title: Periodontal Regeneration of Chronic Periodontal Disease Patients Receiving Stem Cells Injection Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Songlin Wang (Other)
Responsible Party: Sponsor-Investigator, Songlin Wang, Professor and Vice President of Capital Medical University, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CapitalMedicalU-1
Record Dates: First submitted 2015-06-10; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Periodontal Diseases
Keywords: Periodontal Diseases; Bone Regeneration; Dental Pulp Stem Cell
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DPSC injection (Experimental): 20 patients will receive DPSC injection（1000000 cells/ 0.5ml） at the local periodontal defects immediately after periodontal scaling and root planing.
  Interventions: Genetic: DPSC injection
- Placebo control (Placebo Comparator): 20 patients will receive saline injection at the local periodontal defects immediately after periodontal scaling and root planing.
  Interventions: Other: Placebo

INTERVENTIONS:
Genetic: DPSC injection — A 0.5ml saline preparation containing 1000000 DPSCs were injected at the local periodontal defects immediately after periodontal scaling and root planing.
  Arms: DPSC injection
Other: Placebo — A 0.5ml saline preparation were injected at the local periodontal defects immediately after periodontal scaling and root planing.
  Arms: Placebo control

SUMMARY:
The purpose of this study is to evaluate the safety of clinical injection of allogeneic human dental pulp stem cell(DPSC) in local infected periodontal tissue and determine whether injection of allogeneic DPSC is a effective way in the treatment of chronic periodontal disease.

DETAILED DESCRIPTION:
This study will involve 40 patients who were diagnosed as chronic periodontitis will receive periodontal scaling and root planing. Patients will randomly be divided at the base line into two groups.In test group, 20 chronic periodontitis patients will be treated using local DPSC injection. Whereas, a control group will contain 20 patients who will be treated using placebo. Clinical examination including Quigley-Hein plaque index (QHI), bleeding on probing (BoP), probing depth (PD), clinical attachment level (CAL), and gingival recession (GR) will be perform in different time points during the study. Radiographic and clinical examination will be carried out during the late healing phase up to 12 months post operation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of periodontal disease will be based on clinical assessment of:

  * Quigley-Hein index (QHI)
  * Bleeding on Probing (BoP)
  * Pocket Probing Depth (PD)
  * gingival recession (GR)
  * Clinical Attachment Level (CAL)
  * furcation involvement,and
  * radiographical assessment. All patients at the base line of this study should have been received the initial treatment and reached the qualified level of oral hygiene to be included in the next stage.

Exclusion Criteria:

* Pregnant,
* smokers,
* immunosuppressed or diabetes patients,
* patients exhibit gingival hypertrophy,
* require premedication, and
* who have been taking systemic anti-inflammatory medications, or
* have taken antibiotics or
* received periodontal instrumentation within 6 months prior to the study, will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline alveolar bone volume examined by computed tomography(CT) at 1 year | Baseline and 1 year after intervention.

SECONDARY OUTCOMES:
Quigley-Hein plaque index (QHI) | Baseline
Change from Baseline Bleeding on probing (BoP) at 1 year | Baseline and 1 year after intervention.
Change from Baseline Probing depth (PD) at 1 year | Baseline and 1 year after intervention.
Change from Baseline Clinical attachment level (CAL) at 1 year | Baseline and 1 year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Songlin Wang, Ph.D, Study Director — Beijing Key Laboratory of Tooth Regeneration and Function Reconstruction， Capital Medical University School of Stomatology
Locations (1):
- Capital Medical University School of Stomatology, Beijing, Beijing Municipality, China